CLINICAL TRIAL: NCT06831019
Title: The ROAR Study: Reactive Oxygen Species and Reproduction
Acronym: ROAR
Status: Not yet recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 24-42357
Record Dates: First submitted 2025-02-13; First posted 2025-02-17 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Ovarian Aging; IVF Outcome; Oxidative Stress
Keywords: oxidative stress; ovarian aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Follicular fluid, seminal plasma, blood - serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Couples undergoing IVF: Heterosexual couples undergoing IVF
  Interventions: Diagnostic Test: Oxidative stress markers

INTERVENTIONS:
Diagnostic Test: Oxidative stress markers — We will measure markers of oxidative stress in the follicular fluid, semen, and blood and correlate this with IVF and reproductive outcomes

SUMMARY:
This is a prospective cohort study characterizing follicular fluid and serum levels of oxidative stress in women with various infertility diagnoses undergoing in vitro fertilization, and assessing the relationship of oxidative stress to oocyte competence as determined by embryo development outcomes. Furthermore, we will measure oxidative stress in sperm and correlate the overall oxidative stress within the couple with IVF and pregnancy outcomes of the resultant embryos.

ELIGIBILITY:
Inclusion Criteria:

1. Female age 18-43 years
2. Subjects planning blastocyst culture for preimplantation genetic screening (PGS) for aneuploidy.
3. Male partners 18 years of age or older.
4. Must be a registered patient at UCSF Center for Reproductive Health
5. Patient and partner must both be physically present on the day of retreival

Exclusion Criteria:

1. Female partner age 44 or older
2. Planning fresh transfer (hybrid PGS cycle)
3. Cleavage stage biopsy
4. Planning to use frozen sperm

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male and Female couples
Study Population: Heterosexual couples undergoing fresh IVF cycle
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Implantation rate | From enrollment to transfer of all embryos - can be anywhere from 8 weeks to 1 year (or sometimes longer if pregnancy is achieved)
  Implantation rate of euploid embryos that result from a specific oxidative stress environment

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Rosen, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No